CLINICAL TRIAL: NCT02840656
Title: Comparative Microbial Epidemiology and Chlorhexidine Suscebtibily of Oropharyngeal and Intestinal Colonization of Healthy Adults Subjects
Brief Title: Microbial Epidemiology and Chlorhexidine Suscebtibily of Oropharyngeal and Intestinal Colonization
Acronym: OroColi-HS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P140907
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Oropharyngeal Gram-negative Bacilli Colonization

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy adult subject: oropharyngeal and rectal swabbing to collect Gram-negative bacilli
  Interventions: Other: oropharyngeal swabbing; Other: rectal swabbing

INTERVENTIONS:
Other: oropharyngeal swabbing — microbiological sampling will be performed on buccal mucosa with standard swab. only one sample will be done
Other: rectal swabbing — same process as oropharyngeal swabbing will be used to collect rectal microbiological sample

SUMMARY:
In this prospective observational study we aim to determine the prevalence of oropharyngeal and rectal Gram-negative bacilli colonization in healthy subjects, and their susceptibility to chlorehexidine. We plan to recruit 100 healthy volunteers secondary endpoints are to determine the phylogentic characteristics of E. coli isolates; to compare the phylogentic characteristics of oropharyngeal and rectal of predominant GNB colonization.

DETAILED DESCRIPTION:
In this prospective observational study we aim to determine the prevalence of oropharyngeal and rectal Gram-negative bacilli colonization in 100 healthy subjects, and their susceptibility to chlorehexidine. Each participant will undego a oropharyngeal swab collection and a rectal swab at day 0. The Gram-negative bacilli colonization will be identified, E. coli isolates will be studied in terms of phylogeny; gram-negative isolates will be studied in terms of antimicrobial and chlorhexidine susceptibility. The primary objective is to determine the prevalence of oropharyngeal Gram-negative bacilli colonization. The secondary objectives are to determine the chlorhexidine and antimicrobial susceptibility of such colonization; to determine the phylogentic characteristics of oropharyngeal and rectal predominant E. coli isolates; to compare the phylogentic characteristics of oropharyngeal and rectal E. coli isolates.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 yo
* personal history of neck or face irradiation
* no history of gastrointestinal disease
* no symptoms of immunosuppression
* no antibiotic therapy in the previous month
* no hospitalization in the 3 months preceding inclusion
* medical exmination prior to inclusion

Exclusion Criteria:

* affiliated to the social security
* The refusal of a patient to participate in a study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volonteers
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-09; Primary Completion 2017-08-16 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
proportion of patients with an oropharyngeal gram-negative colonization | Day 1

SECONDARY OUTCOMES:
incidence of the a GNB oropharyngeal colonization | Day 1
comparision of the predominant fecal flora with GNB oropharyngeal colonization | Day 1
characterization of antimicrobial and chlorhexidine susceptibility of Gram negative bacteria from oropharyngeal colonization | Day 1
phylogenetic and virulence factor content of E. coli oropharyngeal and rectal colonization | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan MESSIKA, MD, Principal Investigator — Hopital Louis Mourier - Assistance Publique Hopitaux de Paris
Locations (1):
- AP-HP, Louis Mourier Hospital, Colombes, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided